CLINICAL TRIAL: NCT00505726
Title: Reflectance Confocal Imaging of Cervical Intraepithelial Neoplasia (CIN)
Brief Title: Reflectance Confocal Imaging in Cervical Cancer Patients
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ID01-555; CA82880
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Cervical Cancer
Keywords: Cervical Intraepithelial Neoplasia; Cervical Cancer; Reflectance Confocal Imaging; Colposcopy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Confocal Microscopy
  Interventions: Procedure: Reflectance Confocal Imaging

INTERVENTIONS:
Procedure: Reflectance Confocal Imaging — Microscopic images taken during routine colposcopy where disinfected probe inserted into vagina and placed against cervix, 1-3 regions imaged (2 abnormal and one normal), and each taking about 1-2 minutes.

SUMMARY:
The goal of this clinical research study is to see if reflectance confocal microscopy works as well as standard methods to detect cancer of the cervix or precancerous lesions.

Primary Objectives:

1. To identify potential clinical advantages for a noninvasive method of diagnosing dysplasia and neoplasia in the cervix using reflectance confocal microscopy.
2. To obtain real time reflected light images in vivo of sites in the human cervix.
3. To access the effects of acetic acid as a contrast agent for in vivo reflectance confocal imaging.
4. Evaluate the depth of penetration for the fiber optic confocal device and analyze the diagnostic value of images taken from different depths.
5. Determine the sensitivity and specificity of this device for the diagnosis of CIN.

DETAILED DESCRIPTION:
Confocal microscopy may be a new way to detect lesions of the cervix quickly without removing a tissue sample. Women in the study will already be scheduled for colposcopy to detect or treat cervical lesions. (A colposcopy is an exam of the vagina and cervix using a magnifying lens.)

Microscopic images will be taken during the routine colposcopy in the outpatient clinic. A disinfected probe will be inserted into the vagina and placed against the cervix. . The probe sends out laser light and detects reflected light from the tissue. Images of cervical tissue will be formed and displayed on a computer monitor. 1-3 regions of the cervix will be imaged (2 abnormal and one normal), and each will take about 1-2 minutes.

Each imaged site will be biopsied. The biopsies will be analyzed by the research pathologist. The results will be available to participants in the event that care needs to be given. Total participation in this study will be only a few minutes.

This is an investigational study. About 72 women will take part in this study. About 18 will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be individuals 18 years of age or older, who have voluntarily responded to advertisement in the form of posted flyers or word of mouth.
* Subjects must sign an informed consent indicating awareness of the investigational nature of this study.

Exclusion Criteria:

* Pregnant individuals will be ineligible for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women, 18 years of age or older, who are already scheduled for colposcopy to detect or treat cervical lesions.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2001-11; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Reflectance confocal images of cervical tissue in vivo | 1-2 minutes during routine colposcopy

CONTACTS AND LOCATIONS:
Overall Officials: Michele Follen, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- United States (3):
  - Lyndon B. Johnson Hospital, Houston, Texas
  - U. T. Health Science Center, Houston, Texas
  - U.T.M.D. Anderson Cancer Center, Houston, Texas
- British Columbia Cancer Research Center, Vancouver, British Columbia, Canada

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org